CLINICAL TRIAL: NCT05777031
Title: Safety and Efficacy of Collagenase Clostridium Histolyticum After Prior Intralesional Platelet Rich Plasma for Peyronie's Disease
Brief Title: Safety and Efficacy of Collagenase Clostridium Histolyticum After Prior Intralesional PRP for Peyronie's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Thomas Masterson, Assistant professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20221234
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Peyronie Disease; Sexual Dysfunctions, Psychological; Genital Diseases, Male
MeSH Terms: conditions — Penile Induration; Sexual Dysfunctions, Psychological; Genital Diseases, Male | interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Collagenase Clostridium Histolyticum (CCH) Group (Experimental): There will be 8 total treatments. These will follow the manufacturer protocol of 2 injections 24-72 hours apart (one cycle), followed by a 6-week break. This will total a maximum of 4 cycles.
  Interventions: Drug: Collagenase Clostridium Histolyticum (CCH)

INTERVENTIONS:
Drug: Collagenase Clostridium Histolyticum (CCH) — Injection of intralesional CCH (0.58mg) to the penile plaque at the point of maximal curvature. Second injection of each cycle will be injected 2-3mm apart from the prior injection.
  Other Names: Xiaflex

SUMMARY:
The purpose of this study is to learn about the safety and side effects of intralesional collagenase clostridium histolyticum (CCH) injected into the Peyronies Disease (PD) plaque after receiving prior treatment with intralesional Platelet Rich Plasma (PRP) injections.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to provide written informed consent
2. Have a diagnosis of PD with evidence of stable disease as determined by the investigator
3. Patient must have palpable penile plaque
4. Penile curvature deformity of >30° to <90°
5. Agree to comply with all study related tests/procedures.
6. Prior intralesional platelet rich plasma treatment within the past 18 months and desire secondary treatment of penile curvature

Exclusion Criteria:

1. Previous penile surgery of any kind (except circumcision and condyloma removal), such as penile lengthening, penile cancer surgery, penile plication, grafting, penile prosthesis.
2. Previous intralesional injection therapy with CCH for PD within six months. Patients with failed therapy greater than six months ago may be included.
3. Previous history of priapism or penile fracture
4. PD characterized by a ventral plaque
5. Severe erectile dysfunction as characterized with an IIEF score ≤ 12
6. Hour-glass deformity
7. Unwilling to participate
8. Medically unfit for sexual intercourse as deemed by the principal investigator
9. Patients scheduled to undergo an elective medical procedure during the investigation timeframe that will interfere with autologous PRP injection therapy.
10. Have a serious comorbid illness/condition/behavior that, in the opinion of the investigator, may compromise the safety or compliance of the subject or preclude successful completion of the study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment Related Adverse Events | up to 6 months (post-intervention)
  To determine number of treatment related adverse events. Safety will be evaluated via the incidence of adverse events as assessed by treating physician
Percent change of penile curvature in degrees. | Baseline up to 6 months
  Treatment efficacy of CCH will be assessed via the percentage of participants achieving degree change in penile curvature from baseline. Degree of curvature will be measured using a goniometer with the aid of injection of vasoactive substance into the penis.

SECONDARY OUTCOMES:
Change in Peyronie's Disease Questionnaire (PDQ) sub-domain scores (Psychological and Physical Symptoms, Symptom Bother). | Baseline, 6 months.
  Treatment efficacy will be assessed via the change of participants achieving any decrease in Peyronie's disease Questionnaire (PDQ) sub-domain scoring from baseline. The sub-domains that will be assessed in primary outcome is Psychological and Physical Symptoms and Symptom Bother. PDQ is a validated 15-item questionnaire that assess Psychological and Physical Symptoms, Symptom Bother, and Penile Pain subdomains. The Psychological and Physical Symptoms subdomain is measured from 0 to 24 (most severe symptoms). Symptom Bother subdomain is measured from 0 to 30 (most severe pain).
Changes in International Index of Erectile Function - Erectile Function (IIEF-EF) scores | Baseline, 6 months
  IIEF-EF is a 5-item subdomain self-evaluation questionnaire of erectile function. Each item is scored from 0-5 with the total score ranging from 0-25 with the higher score indicating better erectile function.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Masterson, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami - Desai Sethi Urology Institute, Miami, Florida
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: Undecided